CLINICAL TRIAL: NCT05748535
Title: The Effect of Auricular Vagus Nerve Stimulation on Pain and Pulse Variability in Women With Migraine Disease
Brief Title: Effect of Auricular Vagus Nerve Stimulation in Women With Migraine Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Sule Okur, Lecturer, Physiotherapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21.04.2022/28
Record Dates: First submitted 2023-02-20; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Chronic Migraine, Headache
Keywords: Pulse Rate Variability; Pain
MeSH Terms: conditions — Headache; Pain

STUDY DESIGN:
Intervention Model Description: Individuals were divided into three groups as unilateral left, unilateral right and bilateral ear stimulations.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unilateral Right Ear (Experimental): Auricular vagus nerve stimulation performed through the unilateral right ear.
  Interventions: Device: Auricular Vagus Nerve Stimulation
- Unilateral Left Ear (Experimental): Auricular vagus nerve stimulation performed through the unilateral left ear.
  Interventions: Device: Auricular Vagus Nerve Stimulation
- Bilateral Ear (Experimental): Auricular vagus nerve stimulation performed through the bilateral ear.
  Interventions: Device: Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Auricular Vagus Nerve Stimulation — First of all, the application will be explained to the participants and a signed consent form for the application will be obtained from the individuals. Groups; It will be in the form of Right Ear Stimulation, Left Ear Stimulation and Bilateral Ear Stimulation group. Non-invasive auricular vagus nerve stimulation will be applied to all participants with a VAGUSTIM device, biphasic, frequency 10 Hz, pulse width 300 μs in Modulation mode, and current intensity for 20 minutes for 10 sessions, keeping the current constant at the point where the participant feels the current comfortably. Before and after each application, pulse variability (rmssd, LF/HF, pNN50, LF, HF) and blood pressure measurements will be taken from both the right index finger and left index finger. Before the first session and after the 10th session, pain level will be evaluated with the Numerical Pain Rating Scale, and disability level related to headache will be evaluated with the Headache Impact Test.

SUMMARY:
The aim of the study was to investigate the effectiveness of non-invasive auricular vagus nerve stimulation on pain and pulse variability in women aged 18-55 years with migraine. It is also aimed to see the effects of vagus nerve stimulation from all directions by making pain, pulse, blood pressure and autonomic measurements.

DETAILED DESCRIPTION:
Migraine, a neurological disorder that causes severe disability, is characterized by recurrent moderate to severe attacks associated with vegetative symptoms. Patients with frequent attacks may overuse drugs, which can lead to migraine chronization and headache. In the last decade, neuromodulatory approaches have been developed for the treatment of headaches that do not respond adequately to treatment. Non-invasive neuromodulation techniques are an evolving field in migraine research and treatment. Non-invasive vagus nerve stimulation is one of the non-invasive neuromodulation techniques. Promising findings on vagus nerve stimulation in people with chronic pain, including migraine and cluster headaches, are slowly being recognized. Stimulation of the vagus nerve provides a way of regulating autonomic tone. Auricular vagus nerve stimulation regulates abnormal sympatho-vagal balance while activating the parasympathetic system, including anti-inflammatory pathways (cholinergic anti-inflammatory pathway and hypothalamic-pituitary adrenal axis). It is aimed to evaluate the effect on pain and pulse variability after vagus nerve stimulation in women with migraine disease and to learn how the vagus nerve crosses according to the pulse measurements taken from the right and left index fingers.

ELIGIBILITY:
Inclusion Criteria:

* People between the ages of 18-55 with migraine disease
* Having a definite diagnosis of migraine by a neurologist
* Absence of any orthopedic, neurological, etc. diseases that will prevent physical activity
* Not using drugs continuously except for migraine attacks
* Willingness to participate in the study
* Having signed the informed consent form

Exclusion Criteria:

* Cases do not want to continue the study.
* Not signing the informed consent form
* Being on medication for migraine prophylaxis
* Having a communication problem that does not allow evaluation
* Having a history of additional chronic disease that interferes with physical activity,
* Pregnancy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since migraine is seen approximately 3 times more frequently in women than in men, a study consisting of a female population was planned.
Enrollment: 60 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | 1 month
  The Numerical Pain Rating Scale is a widely used scale that requires the patient to rate their pain on a scale of 0 to 10; 0 indicates no pain and 10 reflects the worst possible pain.
Headache Impact Test (HIT-6) | 1 month
  It is a short questionnaire designed to evaluate migraine pain from the patient's perspective and to track the time lost by the patient due to migraine (work, school, housework, social activities).
Pulse Variability/ Elite HRV Cor Sense Monitor | 1 month
  CorSense HRV monitors are used in this study Elite HRV purchased from the company. Readings will be collected through the Elite HRV app designed for mobile devices. The platform is R-R registered via industry standard, according to the Elite HRV website. ranges and defines 0.04-0.15 Hz waves as LF and 0.15-0.40 Hz waves as HF.
Blood Pressure | 1 month
  Blood pressure is the pressure that the heart creates on the vessel wall as it pumps blood through our body.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahcesehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No